CLINICAL TRIAL: NCT00850395
Title: Non-Interventional Study Of Celsentri® In Treatment Experienced Patients Infected With CCR5 Tropic HIV-1
Brief Title: Non-Interventional Study Of Celsentri® In Treatment Experienced Patients With CCR5-Tropic HIV-Infection
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4001070; CELTROP
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Results first posted 2012-10-15 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: HIV-1
Keywords: HIV-1; non-interventional; CCR-5 tropic virus; therapy experienced patients
MeSH Terms: interventions — Maraviroc

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Non-Interventional
  Interventions: Drug: maraviroc

INTERVENTIONS:
Drug: maraviroc — No intervention; any procedure at the discretion of the treating physician, in line with the SmPC
  Other Names: Selzentry, Celsentri

SUMMARY:
Aim of the study is to gain more knowledge about efficacy of CELSENTRI® in daily clinical practice and obtain information about the quality of life of patients using CELSENTRI®.

DETAILED DESCRIPTION:
Non interventional study, inclusion and exclusion criteria defined by the labelling of Celsentri (Maraviroc).

ELIGIBILITY:
Inclusion Criteria:

HIV-1 infection. CCR-5 tropic virus. Therapy experienced patient,

Exclusion Criteria:

X4 or D/M tropic virus. Therapy-naive patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1 infected, therapy-experienced patients, CCR5-tropic virus,
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2009-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001070&StudyName=Non-Interventional%20Study%20Of%20Celsentri%AE%20In%20Treatment%20Experienced%20Patients%20With%20CCR5-Tropic%20HIV-Infection

RESULTS

PARTICIPANT FLOW:
Groups:
- Maraviroc: Participants who were prescribed maraviroc tablets orally in accordance with Summary of Product Characteristics (SmPC) were observed for a period of up to 12 months or early discontinuation.
Period: Overall Study
Arm/Group | Maraviroc
Started | 79
Completed | 69
Not Completed | 10
Not completed — Death | 1
Not completed — Adverse Event | 1
Not completed — Insufficient clinical response | 3
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Arm/Group | Maraviroc
Number analyzed (Participants) | 79
Age Continuous [Mean (Standard Deviation); unit: years] | 44.1 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 67
Log 10 Transformed Human Immunodeficiency Virus-1 Ribonucleic Acid (HIV-1 RNA) [Mean (Standard Deviation); unit: copies/milliliter (copies/mL)] — Number of participants evaluable for this measure=78.
  copies/milliliter (copies/mL) | 3.01 (1.599)
Cluster of Differentiation 4 (CD4+) Cell Counts [Mean (Standard Deviation); unit: cells/microliter (cells/mcL)] | 458.8 (250.14)
Number of Participants With Centers for Disease Control and Prevention (CDC) Classification [Number; unit: participants] — Participants were classified based on the severity as mild (Category A), moderate (Category B), and severe (Category C).
  participants
    Category A | 31
    Category B | 21
    Category C | 27
Acquired Immune Deficiency Syndrome Clinical Trials Group Symptom Distress Module(SDM) Overall Score [Mean (Standard Deviation); unit: units on a scale] — SDM: 20 items questionnaire, each item rated from 0 to 4, 0=complete absence of symptom and 4=very bothersome symptom. Overall score: sum of scores for each of 20 items of questionnaire, with 0=best health and 80=worst health. A positive change from baseline indicates decline in participant's quality of life. Number of participants evaluable=55.
  units on a scale | 17.37 (14.026)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Log 10 Transformed Human Immunodeficiency Virus-1 Ribonucleic Acid (HIV-1 RNA) at Month 3
Time Frame: Baseline, Month 3
Population: Full Analysis Set (FAS) population included all participants who received at least one dose (including partial doses) of study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Maraviroc
Number analyzed (Participants) | 75
copies/mL | -1.10 (1.530)

2. Primary Outcome: Change From Baseline in Log 10 Transformed Human Immunodeficiency Virus-1 Ribonucleic Acid (HIV-1 RNA) at Month 6
Time Frame: Baseline, Month 6
Population: FAS population included all participants who received at least one dose (including partial doses) of study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Maraviroc
Number analyzed (Participants) | 74
copies/mL | -1.15 (1.579)

3. Primary Outcome: Change From Baseline in Log 10 Transformed Human Immunodeficiency Virus-1 Ribonucleic Acid (HIV-1 RNA) at Month 12
Time Frame: Baseline, Month 12
Population: FAS population included all participants who received at least one dose (including partial doses) of study medication. Missing values were imputed as zero for those participants who either discontinued prematurely before the final visit or had missing baseline measurements.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Maraviroc
Number analyzed (Participants) | 79
copies/mL | -0.95 (1.571)

4. Primary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4+) Cell Counts at Month 3
Time Frame: Baseline, Month 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | Maraviroc
Number analyzed (Participants) | 75
cells/mcL | 74.31 (162.18)

5. Primary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4+) Cell Counts at Month 6
Time Frame: Baseline, Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | Maraviroc
Number analyzed (Participants) | 75
cells/mcL | 91.88 (168.43)

6. Primary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4+) Cell Counts at Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | Maraviroc
Number analyzed (Participants) | 79
cells/mcL | 97.57 (237.70)

7. Primary Outcome: Number of Participants With Centers for Disease Control and Prevention (CDC) Classification at Month 3
Description: Participants were classified based on the severity as mild (Category A), moderate (Category B), and severe (Category C).
Time Frame: Month 3
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 76
participants
  Category A | 31
  Category B | 19
  Category C | 26

8. Primary Outcome: Number of Participants With Centers for Disease Control and Prevention (CDC) Classification at Month 6
Description: Participants were classified based on the severity as mild (Category A), moderate (Category B), and severe (Category C).
Time Frame: Month 6
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 74
participants
  Category A | 31
  Category B | 16
  Category C | 27

9. Primary Outcome: Number of Participants With Centers for Disease Control and Prevention (CDC) Classification at Month 12
Description: Participants were classified based on the severity as mild (Category A), moderate (Category B), and severe (Category C).
Time Frame: Month 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 79
participants
  Category A | 31
  Category B | 20
  Category C | 28

10. Secondary Outcome: Change From Baseline in Acquired Immune Deficiency Syndrome (AIDS) Clinical Trials Group (ACTG) Symptom Distress Module (SDM) Overall Score at Months 6 and 12
Description: SDM consists of the 20 items questionnaire, each item rated from 0 to 4 where 0 (complete absence of symptom) and 4 (very bothersome symptom). Overall score calculated as the sum of the scores for each of the 20 items of the questionnaire and ranged from 0 (best health) and 80 (worst health). A positive change from baseline indicates a decline in a participant's quality of life over that period.
Time Frame: Baseline, Months 6, 12
Population: FAS population. 'N' (number of participants analyzed) signifies participants evaluable for this measure. 'n' signifies participants evaluable at specified time point. Missing values were imputed only for Month 12 as zero for those participants who either discontinued prematurely before the final visit or had missing baseline measurements.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maraviroc
Number analyzed (Participants) | 79
units on a scale
  Change at Month 6 (n=51) | -4.87 (12.527)
  Change at Month 12 (n=79) | -2.14 (11.728)

11. Secondary Outcome: Number of Participants With Human Immunodeficiency Virus (HIV) Response
Description: Response was defined as a HIV-1 RNA count of less than 50 copies/mL.
Time Frame: Month 12
Population: FAS population included all participants who received at least one dose (including partial doses) of study medication.
Measure: Number; unit: participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 79
participants | 51

12. Secondary Outcome: Physician's Assessment of Efficacy
Description: Number of participants with each grade of efficacy as assessed by the physician was reported on the 5 point categorical scale: excellent, very good, good, fair, poor.
Time Frame: Month 12
Population: FAS population included all participants who received at least one dose (including partial doses) of study medication.
Measure: Number; unit: participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 79
participants
  Excellent | 15
  Very Good | 42
  Good | 14
  Fair | 1
  Poor | 1

13. Secondary Outcome: Number of Participants Taking Concomitant Therapy
Description: Participants taking HIV/AIDS concomitant medication at Month 12, at Baseline and Month 12 were reported. It included Emtricitabine/tenofovir disoproxil fumarate(FTC/TDF),Raltegravir(RAL), Ritonavir (RTV), Darunavir(DRV), Kaletra, Atazanavir sulfate(ATV), Abacavir sulfate/lamivudine(ABC/LAM), Tenofovir disoproxil fumarate(TDF), Etravirine(ETR), Lamivudine (LAM), Zidovudine W/lamivudine(ZDV W/LAM), Nevirapine(NVP), Saquinavir mesilate(SQV), Trizivir(TZV), Zidovudine(ZDV), Abacavir sulfate(ABC), Emtricitabine(FTC),Entecavir(ETV).
Time Frame: Baseline, Month 12
Population: FAS population included all participants who received at least one dose (including partial doses) of study medication.
Measure: Number; unit: participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 79
participants
  ABC, FTC/TDF (Month 12) | 1
  ABC, FTC/TDF (Baseline, Month 12) | 1
  ABC/LAM (Month 12) | 2
  ABC/LAM (Baseline, Month 12) | 2
  ABC/LAM, DRV, RAL (Month 12) | 1
  ABC/LAM, DRV, RAL (Baseline, Month 12) | 0
  ABC/LAM, RAL (Month 12) | 2
  ABC/LAM, RAL (Baseline, Month 12) | 2
  ABC/LAM, RAL, TDF (Month 12) | 1
  ABC/LAM, RAL, TDF (Baseline, Month 12) | 1
  ATV (Month 12) | 1
  ATV (Baseline, Month 12) | 1
  ATV, FTC/TDF (Month 12) | 1
  ATV, FTC/TDF (Baseline, Month 12) | 1
  ATV, FTC/TDF, RTV (Month 12) | 1
  ATV, FTC/TDF, RTV (Baseline, Month 12) | 1
  ATV, LAM, RAL, RTV (Month 12) | 1
  ATV, LAM, RAL, RTV (Baseline, Month 12) | 0
  ATV, RAL (Month 12) | 2
  ATV, RAL (Baseline, Month 12) | 2
  ATV, RAL, RTV (Month 12) | 1
  ATV, RAL, RTV (Baseline, Month 12) | 1
  ATV, RTV (Month 12) | 1
  ATV, RTV (Baseline, Month 12) | 1
  DRV, FTC/TDF (Month 12) | 1
  DRV, FTC/TDF (Baseline, Month 12) | 1
  DRV, FTC/TDF, ETR (Month 12) | 1
  DRV, FTC/TDF, ETR (Baseline, Month 12) | 1
  DRV, FTC/TDF, RTV (Month 12) | 6
  DRV, FTC/TDF, RTV (Baseline, Month 12) | 5
  DRV, ETV, ETR, RTV (Month 12) | 1
  DRV, ETV, ETR, RTV (Baseline, Month 12) | 0
  DRV, LAM, RAL (Month 12) | 1
  DRV, LAM, RAL (Baseline, Month 12) | 0
  DRV, LAM, RAL, RTV (Month 12) | 1
  DRV, LAM, RAL, RTV (Baseline, Month 12) | 0
  DRV, LAM, TDF (Month 12) | 1
  DRV, LAM, TDF (Baseline, Month 12) | 1
  DRV, NVP, RAL, RTV (Month 12) | 1
  DRV, NVP, RAL, RTV (Baseline, Month 12) | 1
  DRV, RAL, RTV (Month 12) | 4
  DRV, RAL, RTV (Baseline, Month 12) | 4
  DRV, RTV (Month 12) | 2
  DRV, RTV (Baseline, Month 12) | 2
  DRV, RTV, TZV (Month 12) | 1
  DRV, RTV, TZV (Baseline, Month 12) | 1
  FTC/TDF (Month 12) | 13
  FTC/TDF (Baseline, Month 12) | 11
  FTC/TDF, Kaletra (Month 12) | 2
  FTC/TDF, Kaletra (Baseline, Month 12) | 1
  FTC/TDF, Kaletra, RAL (Month 12) | 3
  FTC/TDF, Kaletra, RAL (Baseline, Month 12) | 3
  FTC/TDF, Kaletra, SQV (Month 12) | 1
  FTC/TDF, Kaletra, SQV (Baseline, Month 12) | 1
  FTC/TDF, RAL (Month 12) | 5
  FTC/TDF, RAL (Baseline, Month 12) | 4
  FTC/TDF, RAL, SQV (Month 12) | 1
  FTC/TDF, RAL, SQV (Baseline, Month 12) | 1
  ETR, RAL, RTV (Month 12) | 1
  ETR, RAL, RTV (Baseline, Month 12) | 0
  Kaletra (Month 12) | 2
  Kaletra (Baseline, Month 12) | 2
  LAM, RAL, TDF, ZDV (Month 12) | 1
  LAM, RAL, TDF, ZDV (Baseline, Month 12) | 0
  RAL (Month 12) | 2
  RAL (Baseline, Month 12) | 2
  RAL, TDF (Month 12) | 1
  RAL, TDF (Baseline, Month 12) | 1
  RAL, ZDV W/LAM (Month 12) | 1
  RAL, ZDV W/LAM (Baseline, Month 12) | 1
  TDF, TZV (Month 12) | 1
  TDF, TZV (Baseline, Month 12) | 1
  TDF, ZDV (Month 12) | 1
  TDF, ZDV (Baseline, Month 12) | 1

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Maraviroc
Serious Adverse Events (participants affected / at risk) | 3/79
Other Adverse Events (participants affected / at risk) | 4/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc (N=79)
Ichthyosis (Congenital, familial and genetic disorders) | 1
Pneumonia (Infections and infestations) | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Suicide attempt (Psychiatric disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc (N=79)
Bronchitis (Infections and infestations) | 4

LIMITATIONS AND CAVEATS:
Designation of outcomes as primary and secondary was based on study team input as study did not specify primary or secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.